CLINICAL TRIAL: NCT06582212
Title: Enabling Women with Parkinson's Disease to Identify and Better Manage Hormonal Triggers
Brief Title: Enabling Women with Parkinson's Disease to Identify and Better Manage Hormonal Triggers of Parkinsonian Symptoms
Acronym: Lady-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC24.0082; 2024-A00598-39 (Other: ID RCB)
Record Dates: First submitted 2024-06-24; First posted 2024-09-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Digital Technology; Mobile Application; Motor Fluctuations; Oestrogen; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MyMovesMatter mobile application (Experimental)
  Interventions: Device: Mymovesmatter mobile application

INTERVENTIONS:
Device: Mymovesmatter mobile application — Patients with Parkinson's disease will use a mobile application (Mymovesmatter) to evaluate changes in motor and non motor symptoms during their hormonal cycles.

SUMMARY:
Forty percent of people living worldwide with Parkinson's disease (PD) are women. Twenty percent of patients have PD onset under the age of 60 years, a time when women may encounter significant caregiving responsibilities along with occupational and other competing demands.

Studies with surveys of women with PD (WwPD) have reported worsening of PDrelated symptoms especially in the week prior and the week of menses. However, prospective evidence is scarce and clinical guidelines to manage this issue do not exist. As a result, care is either non-existent or fragmented.

The investigators propose a French multicentre prospective pilot study to capture changes in PD symptoms in relation to the stages of the menstrual cycle aiming at reducing hormonal related worsening in PD symptoms through neurologist intervention and/or patient selfmanagement.

Digital technology will remotely enable patient reported outcome (PRO) tracking through the My Moves Matter app changes in PD symptoms during several months. This information will then help neurologists to customize treatment.

Changes in motor symptoms will also be highlighted by tracking through the use of a wearable device (PDMonitor) to objectively detect motor changes together with the app.

This will further support the reliability of the app. This study will provide evidence for the impact of the menstrual cycle on PD and help neurologists and patients to better manage PD symptoms related to these hormonal changes.

DETAILED DESCRIPTION:
This is a prospective multicentre pilot study of the impact of the menstrual/hormonal cycle on PD symptoms and their treatment in pre-menopausal WwPD based on the remote tracking of PD symptoms and menstrual/hormonal cycle through the MMM digital health app in the French language.

There is an ongoing European preliminary study investigating the usability of the MMM App to track menstrual symptoms in WwPD, endorsed by the Parkinson's Disease Research Cluster in the University College Cork in Ireland.

The aim of that study does not overlap with the current proposal.

The aims of the LADY-PD project are:

1. Aim 1. To determine the reliability of using our new mobile application to track motor and non-motor symptoms in pre-menopausal WwPD. French WwPD will use the My Moves Matter (MMM) application downloaded in their mobile phone to track their PD symptoms during their hormonal cycle. Changes during the cycle can be identified using a linear system to quantify changes in each symptom. The investigators will measure drop-out rate, missing data, usability, and acceptability (the latter with questionnaires for patients and neurologists).
2. Aim 2. To compare the mobile application subjective motor data against the gold standard clinical scale, the motor part of the Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS). This will be done acquiring data coming from a subset of WwPD who will have an objective measurement of the MDS-UPDRS (using the PDMonitor, a digital device able to measure bradykinesia, tremor, gait, posture, rigidity, dyskinesia) while using the mobile application.

   Statistical analysis will compare data between the two devices.
3. Aim 3. To determine the clinical efficacy of interventions (changes on medication, physiotherapy, et cetera) suggested by the neurologists to improve motor and nonmotor symptoms detected by the mobile application during the initial 3-month period of evaluation. Effects of pharmacological and non-pharmacological interventions will be measured using the mobile app after a 3-month period of evaluation.

The investigators hypothesize that

1. pre-menopausal WwPD will experience a worsening of motor and NMS during their menstrual/hormonal cycle (and possibly independently by OCP treatment);
2. these changes will have a relevant impact on the well-being of patients, and on their daily and social activities;
3. appropriate management of these changes can effectively improve quality of life of pre-menopausal WwPD.

ELIGIBILITY:
Inclusion Criteria:

* Non-menopausal women
* Diagnosis of PD according to the MDS criteria onset of PD symptoms since at least two years before inclusion
* Age 18-56 years
* On stable medication regimen for PD for at least two months without foreseen need to modify it within the next three months
* With and without OCP or intrauterine devices (IUD

Exclusion Criteria:

* Post-menopausal women with PD
* Any condition that, in the opinion of the investigator, will preclude the participant from successfully or safely completing study procedures (i.e., dementia, severe depression, etc.)
* People not able to give an informed consent.

Ages: 18 Years to 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-03-12 (Estimated); Study Completion 2027-09-12 (Estimated)

PRIMARY OUTCOMES:
Reliability of the MyMovesMatter mobile application | Inclusion, 3 months and 6 months
  Changes in PD symptoms collected during the menstrual/hormonal cycle versus those collected in the other days of the month. These changes will be evaluated using a linear system included in the My Moves Matter application. In particular, bradykinesia, tremor, gait, posture, dyskinesia, fatigue, anxiety, pain, urinary disturbances and sweating will be assessed.

SECONDARY OUTCOMES:
Subjective versus objective evaluation of Parkinson's disease symptoms | Inclusion, 3 months and 6 months
  Subjective motor variables obtained with the mobile application will be compared to the the gold standard clinical scale, the related items Movement Disorders Society -Unified Parkinson Disease Rating Scale part III (0-132) and IV (0-24). Lower scores mean a better outcome.
To determine the clinical efficacy of interventions | At 3 months and 6 months
  Clinical efficacy of interventions suggested by the neurologists to improve motor and non-motor symptoms detected by the mobile application during the initial 3-month period of evaluation will be evaluated by analysing the scores' differences between T1 and T2 using the My Moves Matter application.
To evaluate whether Woman with Parkinson's disease with and without contraception have different clinical outcomes | Inclusion, 3 months and 6 months
  To evaluate whether Woman with Parkinson's disease with and without contraception have different clinical outcomes.
  The total sample will be divided into two sub-groups (with vs. without contraception) and the effect of Period will be compared between the two sub-groups using ANOVA (GLM) for repeated measures, with Group as an inter-subjects' factor and Period as an intra-subject factor.
Usability of the system | At 6 months
  Usability of the system will be examined using the System Usability Scale score (max 100) averaged across participants. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elena MORO, Principal Investigator — CHU Grenoble Alpes
Locations (4):
- France (4):
  - CHU Grenoble Alpes, Grenoble, Grenoble
  - CHU Nantes Hôpital Laennec, Nantes
  - CHU Rennes -Site Pontchaillou, Rennes
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No